CLINICAL TRIAL: NCT06786221
Title: Accuracy, Stability and Safety of Orthodontic Mini-implant Template in the Infrazygomatic Crest Zone
Acronym: CAD/CAM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Su li, phd, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Beijing Xuanwu Tcm Hospital; XWKX2024-32 (Other Grant/Funding Number: Beijing Xicheng District Health Commission)
Record Dates: First submitted 2024-11-20; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Dental Implants; Dental Implantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mini-implant template (Experimental): Participants in this arm will undergo micro-implant surgery using a digitally designed and 3D-printed micro-implant guide template.
  Details:
  The guide template is created based on preoperative CT scans of the participant's anatomy.
  The template is used during the surgery to precisely guide the placement of micro-implants in terms of position, angle, and depth.
  The surgery is performed with the assistance of the digital guide to ensure accuracy and reduce the risk of complications.
  Data on the stability of the guide, implant accuracy, and surgical time are recorded.
  Interventions: Device: mini-implant template
- Control Group (No Intervention): Participants in this arm will undergo traditional freehand micro-implant surgery without the use of any guide template or digital assistance.
  Details:
  The surgery relies entirely on the surgeon's experience and manual operation. No digital or physical guides are used during the procedure. Data on surgical time, implant accuracy, and any post-operative complications are recorded.
  This arm serves as the control group to compare the outcomes with those of the experimental group.

INTERVENTIONS:
Device: mini-implant template — The proposed structure will be made of three main components: a tooth guide part, a gingival guide part, and a steering part. The tooth guide and gingival guide parts are firmly connected by fracture lines. The mini-implant guide part is specifically designed to accommodate the angle and position required for miniscrew insertion. On the basis of the resin guide plate, add a guide hole structure and change it to simulate the patient's actual tooth root condition.
  During usage, the guide can be pre-designed in accordance with the desired planting position and direction of the patient's mini-implant, enabling precise guidance during the implantation process. The designed guide's data is inputted into EnvisionTEC Vida 3D printer to create the mini-implant guide. Prior to the implantation of the mini-screw, patients will be informed about the potential risks and required to sign an informed consent form.
  Arms: mini-implant template

SUMMARY:
The goal of this clinical trial is to learn accuracy, stability and safety of orthodontic mini-implant template in the infrazygomatic crest zone.References population isOrthodontics patients which is require to implant miniscrew as anchorage requirement .Inclusion criteria

1. The orthodontic clinical design should include the use of miniscrews for anchorage requirements in maxillary arch.
2. Age of 18-35 years old
3. Patients must have no prior history of orthodontic treatment and must have a healthy periodontal condition or no history of trauma before the current orthodontic treatment.

Exclusion criteria

1. Patient with poor oral hygiene, history of systemic diseases and metal allergies;
2. Patients with osteoporosis and inability to retain the TAD;
3. Patients who require orthognathic surgery for severe skeletal malocclusion;
4. Smoking patients which will affect the success rate of the implant placement
5. Patients with incomplete medical records.

The main questions it aims to answer are:

The general objective of this research is to study the effect of utilizing modified miniscrew template as tools for the miniscrew placement.

Specific Objective

The specific objectives for this study will be:

1. To compare the accuracy of miniscrews implanted using modified template by computer-aided design and without template guide (conventional method).
2. To compare the stability of miniscrews implanted using modified template by computer-aided design and without templete guide (conventional method).
3. To compare the safety of miniscrews implanted using modified template by computer-aided design and without templete guide (conventional method).

Participants will:

1. The patient undergoes routine pre-orthodontic examination, model analysis, cephalometric measurement, and develops an orthodontic treatment plan.
2. .The patient undergoes routine pre-orthodontic examination, model analysis, cephalometric measurement, and develops an orthodontic treatment plan.
3. The process of insertion of miniscrew will be depend on the group either Intervention Group or Control Group. The guide plate will be used for miniscrew insertion in Intervention Group and experience based on the patient's digital films for Control Group. The area of insertion of the miniscew will be the upper alveolar ridge between premolars and molar tooth. The procedure will be performed under local injection anesthesia.
4. The process of implanting implant nails on Intervention Group is as follows: the material and model of the implanted micro implant nails are exactly the same as those of the traditional positioning set. The implant nail diameter is 2mm and the length is 10 mm. The implant surgery was performed by the same orthodontist in accordance with recommended operating procedures. Preoperative local anesthesia will be performed, and micro-implant nails will be implanted at the intended implantation site under the guidance of the guide plate. The area of implantation is maxillary zygomatic alveolar ridge.

5）The process of implanting implant nails on the Control Group is as follows: Similar to the intervention group, but the doctor implant the miniscrew based on experience with CBCT scans.

6) Collect date before and after implant nail implantation.The digital plaster models will be obtained by scanning with a D700 scanner (3shape, Denmark). Both digital models and CBCT scan data will be imported into Segma implant guide software (Beijing, China). The combination method is as follows: first, open the file in a way that only uses CBCT for implant design and adjust the density of anatomical landmarks such as the maxillary sinus, condylar foramen, or protrusions to an explicit level. Then, the teeth or jaw landmark points of the model and CBCT will be selected to reconstruct a 3D model.

4）The data collection will be performed by obtaining plaster model using intaoral scanner at T1(immediate post insertion) and T2 (6 months post insertion)

ELIGIBILITY:
Inclusion Criteria:

* The orthodontic clinical design should include the use of miniscrews for anchorage requirements in maxillary arch.
* Age of 18-35 years old.
* Patients must have no prior history of orthodontic treatment and must have a healthy periodontal condition or no history of trauma before the current orthodontic treatment.

Exclusion Criteria:

* Patient with poor oral hygiene, history of systemic diseases and metal allergies.
* Patients with osteoporosis and inability to retain the TAD.
* Patients who require orthognathic surgery for severe skeletal malocclusion.
* Smoking patients which will affect the success rate of the implant placement.
* Patients with incomplete medical records.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Implant Placement | up to 6 months
  The primary goal is to assess the accuracy of implant placement using the orthodontic mini-implant template in the infrazygomatic crest zone. This will be measured by comparing the planned implant position (based on preoperative imaging) with the actual implant position achieved during surgery.
Stability of Implant | up to 6 months
  The stability of the mini-implants will be assessed to ensure they remain securely in place during the orthodontic treatment period.
Safety and Adverse Events | up to 6 months
  e safety of the mini-implant template will be evaluated by recording any adverse events or complications related to the implant surgery or the use of the template.

CONTACTS AND LOCATIONS:
Overall Officials: Norma Ab Rahman, phd, Study Director — Universiti Sains Malaysia
Locations (1):
- Beijing Xuanwu Tcm Hospital, Beijing, Beiijng, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

DOCUMENTS (2):
  • Study Protocol (2024-12-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT06786221/Prot_000.pdf
  • Informed Consent Form (2024-12-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT06786221/ICF_001.pdf